CLINICAL TRIAL: NCT03119194
Title: An Open-Label, Single-Dose, Single-Period Study Designed to Assess the Mass Balance Recovery, Metabolite Profile and Metabolite Identification of [14C]-BIA 9-1067 in Healthy Male Subjects
Brief Title: Mass Balance Recovery, Metabolite Profile and Metabolite Identification of [14C]-BIA 9-1067
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BIA-91067-130
Record Dates: First submitted 2017-04-13; First posted 2017-04-18 (Actual); Last update posted 2017-08-24 (Actual); Status verified 2017-08

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Reguimen A - [14C]-BIA 9-1067 (Experimental): 100 mg [14C]-BIA 9-1067 Capsule containing not more than 3.3 MBq (89.2 µCi) 14C; will be administered with 240 mL water.
  Single dose administration on a single occasion.
  Interventions: Drug: [14C]-BIA 9-1067

INTERVENTIONS:
Drug: [14C]-BIA 9-1067 — 1 × 100 mg capsule, Oral

SUMMARY:
The purpose is to and to assess the mass balance recovery after a single oral dose of [14C]-BIA 9-1067 and to provide plasma, urine and faecal samples for metabolite profiling and structural identification.

DETAILED DESCRIPTION:
This is an open-label, single-dose, single-period, non-randomised study in healthy male subjects. Subjects will be screened for eligibility to participate in the study between 28 and 2 days before dosing. Eligible subjects will be admitted to the clinical unit on the evening of the day before dosing (Day -1). Subjects will be dosed on the morning of Day 1 following an overnight fast of approximately 8 h. Blood, urine, faeces and expired air will be collected at predefined time points for mass balance and PK analysis. Subjects will remain resident in the clinic until the morning of Day 22, when they will be discharged as a group.

Single dose administration on a single occasion. The estimated duration of the study from screening until the final return visit is approximately 3.5 months.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males;
* Age 30 to 65 years of age;
* Body mass index of 18.0 to 35.0 kg/m2 or, if outside the range, considered not clinically significant by the investigator;
* Normal resting supine blood pressure and pulse or showing no clinically relevant deviation as judged by the investigator;
* Computerized (12-lead) ECG recording without signs of clinically relevant pathology or showing no clinically relevant deviations as judged by the investigator;
* All values for clinical laboratory tests of blood and urine within the normal range or showing no clinically relevant deviations as judged by the investigator;
* Must be willing and able to communicate and participate in the whole study;
* Must have regular bowel movements (i.e. average stool production of ≥1 and ≤3 stools per day);
* Must provide written informed consent;
* Must agree to use an adequate method of contraception

Exclusion Criteria:

* Females;
* Subjects who have received any IMP in a clinical research study within the previous 3 months;
* Subjects who are study site employees, or immediate family members of a study site or sponsor employee;
* Subjects who have previously been enrolled in this study;
* History of any drug or alcohol abuse in the past 2 years;
* Regular alcohol consumption in males >21 units per week (1 unit = ½ pint beer, 25 mL of 40% spirit or a 125 mL glass of wine);
* Current smokers and those who have smoked within the last 12 months. A breath carbon monoxide reading of greater than 10 ppm at screening and admission;
* Current users of e-cigarettes and nicotine replacement products and those who have used these products within the last 12 months
* Radiation exposure, including that from the present study, excluding background radiation but including diagnostic x-rays and other medical exposures, exceeding 5 mSv in the last 12 months or 10 mSv in the last 5 years. No occupationally exposed worker, as defined in the Ionising Radiation Regulations 1999, shall participate in the study;
* Subjects who do not have suitable veins for multiple venepunctures/cannulation as assessed by the investigator at screening;
* Clinically significant abnormal biochemistry, haematology or urinalysis as judged by the investigator;
* Positive drugs of abuse test result;
* Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) or human immunodeficiency virus (HIV) results;
* Evidence of renal impairment at screening, as indicated by an estimated creatinine clearance of <90 mL/min using the Cockcroft-Gault equation;
* History of cardiovascular, neurological, renal, hepatic, chronic respiratory or gastrointestinal disease, or clinically significant psychiatric history as judged by the investigator;
* Serious adverse reaction or serious hypersensitivity to any drug or the formulation excipients
* Presence or history of clinically significant allergy requiring treatment, as judged by the investigator. Hayfever is allowed unless it is active;
* Donation or loss of greater than 400 mL of blood within the previous 3 months;
* Subjects who are taking, or have taken, any prescribed or over-the-counter drug (other than 2 g per day paracetamol) or herbal remedies in the 14 days before IMP administration. Exceptions may apply on a case by case basis, if considered not to interfere with the objectives of the study, as agreed by the PI and sponsor's medical monitor;
* Failure to satisfy the investigator of fitness to participate for any other reason.

Ages: 30 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2017-01-27 (Actual); Primary Completion 2017-04-27 (Actual); Study Completion 2017-04-27 (Actual)

PRIMARY OUTCOMES:
Mass balance recovery of total radioactivity in all (urine, faeces and expired air combined) amount excreted (Ae) expressed as a percentage of the administered dose (%Ae) | Urine and faeces: pre-dose,0,0.25,0.5,0.75,1,1.5, 2, 3, 4, 6,8,12,18,24,36,48,72,96,120,144,168,240,312,408,504,648 hours after dosing. Expired air: Pre-dose, 0.5,1,1.5,2,4,6,8,12,18,24,36,48,72,96,120,168,240,312,408,504 hours after dosing.
  Mass balance of total radioactivity in urine, faeces and expired air
Mass balance recovery of total radioactivity in all (urine, faeces and expired air combined) cumulative recovery (CumAe) expressed as a percentage of the administered dose (Cum%Ae) | Urine and faeces: pre-dose,0,0.25,0.5,0.75,1,1.5, 2, 3, 4, 6,8,12,18,24,36,48,72,96,120,144,168,240,312,408,504,648 hours after dosing. Expired air: Pre-dose, 0.5,1,1.5,2,4,6,8,12,18,24,36,48,72,96,120,168,240,312,408,504 hours after dosing.
  Mass balance of total radioactivity in urine, faeces and expired air

SECONDARY OUTCOMES:
Tlag: the elapsed time from dosing at which analyte was first quantifiable in a concentration vs time profile | Pre-dose, 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 120, 240, 408, 504 hours after dosing
  Pharmacokinetic Data Analysis for BIA 9-1067 and its metabolites, BIA 9-1103 and BIA 9-4588
Cmax: maximum observed concentration | Pre-dose, 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 120, 240, 408, 504 hours after dosing
  Pharmacokinetic Data Analysis for BIA 9-1067 and its metabolites, BIA 9-1103 and BIA 9-4588
Tmax: the time from dosing at which Cmax was apparent | Pre-dose, 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 120, 240, 408, 504 hours after dosing
  Pharmacokinetic Data Analysis for BIA 9-1067 and its metabolites, BIA 9-1103 and BIA 9-4588
AUC0-t: area under the curve from 0 time to last measurable concentration | Pre-dose, 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 120, 240, 408, 504 hours after dosing
  Pharmacokinetic Data Analysis for BIA 9-1067 and its metabolites, BIA 9-1103 and BIA 9-4588

CONTACTS AND LOCATIONS:
Locations (1):
- Quotient Clinical, Ruddington, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided